CLINICAL TRIAL: NCT06791291
Title: Efficacy and Safety of Teplizumab in the Treatment of Japanese Pediatric and Adult Participants Aged 8 to 34 Years With Stage 2 Type 1 Diabetes: A Multicenter, Randomized, Open-label, Controlled Study.
Brief Title: Efficacy and Safety of Teplizumab in Japanese Participants With Stage 2 Type 1 Diabetes
Acronym: KIBOU-T1D
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACT18487; U1111-1308-1324 (Registry Identifier: ICTRP); jRCT2031240637 (Registry Identifier: JRCT)
Record Dates: First submitted 2025-01-20; First posted 2025-01-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — teplizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Teplizumab (Experimental): Participants will receive Teplizumab via IV infusion
  Interventions: Drug: Teplizumab
- Control (No Intervention): Participants will receive no treatment in the control group

INTERVENTIONS:
Drug: Teplizumab — Pharmaceutical form:Solution for injection-Route of administration:Intravenous infusion
  Other Names: SAR446681; TZIELD
  Arms: Teplizumab

SUMMARY:
This is a parallel, Phase 2, two-arm study to assess the efficacy and safety of 14-days intravenous (IV) infusion of teplizumab treatment.

Teplizumab has been approved by FDA to delay the onset of Stage 3 Type 1 Diabetes (T1D) in adults and pediatric patients aged 8 years and older with Stage 2 T1D. The dose regimen of teplizumab in this study is consistent with the regimen approved by US FDA.

Given prior clinical studies conducted in Western countries, this design is appropriate to assess the efficacy, safety and tolerability, pharmacokinetic, pharmacodynamic, and immunogenicity of a 14-day IV infusion regimen of teplizumab in Japanese Stage 2 T1D participants aged 8 to 34 years.

DETAILED DESCRIPTION:
Total study duration is approximately 756 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Japanese participant, 8 (inclusive) to 34 years (inclusive) of age, at the time of signing the informed consent. Japanese: born in Japan or ethnic Japanese born outside of Japan, and a descendent of 4 ethnic Japanese grandparents who were all born in Japan.
* Confirmed diagnosis of Stage 2 T1D based on following criteria:
* Participant is positive for 2 or more T1D related auto-antibodies (confirmed by written medical history and/or obtained at study screening). The autoantibodies that are to be confirmed are anti-GAD (glutamic acid decarboxylase), anti-IA2 (insulinoma-associated antigen 2), anti-insulin, anti-ZnT8 (zinc transporter 8), and/or ICA (islet cell antibody).
* Oral glucose tolerance test (OGTT) or blood HbA1c confirms the participant has dysglycemia without overt hyperglycemia.
* Participant must be in good health (except for being Stage 2 T1D) as determined by medical e)valuation including medical history, physical examination, laboratory tests, and electrocardiogram (ECG) XE " ECG " \f Abbreviation \t "electrocardiogram" .
* Participant is up to date with routine age-appropriate immunizations according to current local specific guideline prior to randomization.
* Female participants should use contraceptives consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* A female participant is considered fertile (woman of childbearing potential - WOCBP) from the time of menarche until becoming postmenopausal unless permanently sterile. Female participants are eligible to participate if one of the following conditions applies:
* Is a woman of nonchildbearing potential (WONCBP) OR
* Is a WOCBP and agrees to keep abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent, or use other highly effective contraceptive method, from signing of the informed consent to at least 3 months and 2 weeks after randomization and agrees not to donate or cryopreserve eggs (ova, oocytes) for the purpose of reproduction during this period.

A WOCBP must have at least a negative highly sensitive pregnancy test within 48 hours before the administration of study intervention.

If a urine test cannot be confirmed as negative (eg, an ambiguous result), a blood pregnancy test is required. In such cases, the participant must be excluded from participation if the serum pregnancy result is positive.

Participants are excluded from the study if any of the following criteria apply:

* Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, dermatologic, hepatic, renal, metabolic (except Stage 2 T1D), hematological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, gynecologic (if female), or infectious disease, or signs of acute illness.
* Participant has clinical signs and symptoms consistent with COVID19, eg, fever, dry cough, dyspnea, loss of taste and smell, sore throat, fatigue or confirmed infection by appropriate laboratory test within the last 4 weeks prior to Screening. Participant who had severe course of COVID-19 (ie, hospitalization, extracorporeal membrane oxygenation, mechanically ventilated).
* For participant ≥18 years, blood donation of 400 mL within 12 weeks (male) or 16 weeks (female), 200 mL within 4 weeks or apheresis donation within 2 weeks before randomization; for participant <18 years, blood donation of any volume within 16 weeks before randomization; for any participant, blood transfusion (any volume) within 2 months before randomization.
* Presence or history of drug hypersensitivity to any biologic medication, or clinically significant allergic disease as diagnosed and treated by a physician. Participants with known hypersensitivity to teplizumab or components of the teplizumab injection (including sodium phosphate, sodium chloride, polysorbate 80).
* Participants with a history of active or latent or inactive tuberculosis (TB), including chest X-ray consistent with TB, regardless of treatment, or have a positive QuantiFERON-TB Gold test or T-SPOT TB test at screening.
* At screening, participant has laboratory or clinical evidence of acute or clinically active infection with Epstein Barr virus (EBV), or history of infectious mononucleosis within 3 months before enrollment.
* At screening, participant has laboratory or clinical evidence of acute or clinically active infection with cytomegalovirus (CMV).
* Participants with a history of invasive opportunistic infections, such as histoplasmosis, listeriosis, coccidioidomycosis, candidiasis, pneumonocystis jirovecii, aspergillosis, irrespective of resolution.
* Participants have other autoimmune diseases, except clinically stable autoimmune thyroid disease, or celiac disease.
* Participants with a history of malignancy occurring within 5 years before randomization (except successfully treated carcinoma in situ of the cervix, or adequately treated nonmetastatic squamous cell or basal cell carcinoma of the skin).
* Participants with fever (temperature ≥38.0°C) within 48 hours before randomization; or with chronic persistent or recurring infection(s) requiring active treatment with antibiotics, antiviral or antifungals within 4 weeks before randomization; or with other frequent recurrent infections deemed unacceptable as per Investigator's judgement.
* If female, pregnancy (defined as positive blood or urine pregnancy test) or breast-feeding.
* Participant has recent or planned vaccinations as follows:
* Live vaccines: within 8 weeks before randomization, and/or within 54 weeks after randomization.
* Non-live vaccines: any initial non-live vaccination within 2 weeks before randomization, and/or within 8 weeks after randomization.
* Participant has a current or prior (within 30 days before randomization) treatment that is known to cause a significant, ongoing change in the course of T1D or immunologic status, including high dose, inhaled, extensive topical, or systemic glucocorticoids.
* Participant has a current or prior (within 30 days before randomization) treatment that is known to significantly influence glucose tolerance (anti-hyperglycemic agents, atypical antipsychotics, diphenylhydantoin, niacin etc.).
* Participant has received any anti-CD3 (cluster of differentiation 3) antibody treatment (including teplizumab) before randomization.
* Participant who has received any biologic therapy within five half-lives of the therapy or within 6 months before randomization whichever is longer, or plan to receive any biologic therapy within 6 weeks after randomization.
* Any participant enrolled or having participated, in this or any other clinical study involving an investigational medicinal product (IMP) or in any other type of medical research and is still in the exclusion period according to applicable regulations (eg, having received an IMP of new active pharmaceutical ingredient (API) within 4 months or that of an approved API within 3 months before the administration of this study's IMP).
* Participant has any of the following hematologic parameters before randomization:
* Lymphocyte count <1.0 ×109/L.
* Neutrophil count <1.5 ×109/L.
* Platelet count <150 ×109/L.
* Hemoglobin <100 g/L.
* Participant has any of the following liver function test abnormalities before randomization:
* AST >2 × ULN (upper limit normal).
* ALT >2 × ULN.
* Total bilirubin >1.5 × ULN with the exception of participants with the diagnosis of Gilbert's syndrome who may be eligible provided they have no other causes leading to hyperbilirubinemia.
* Positive result on any of the following tests:
* Hepatitis B surface antigen or hepatitis B core antibody confirmed by positive HBV-DNA (hepatitis B virus DNA).
* Anti-hepatitis C virus antibody confirmed by positive HCV-RNA (hepatitis C virus RNA).
* Human immunodeficiency virus antigen/ antibodies.
* Positive SARS-CoV-2 test.
* Participant who has contraindications or known allergy to both nonsteroidal anti-inflammatory drugs (NSAIDs) and acetaminophen, or anti-histamines and in the opinion of the Investigator, cannot participate in the study.
* Participant not suitable for participation, whatever the reason, as judged by the Investigator, including medical or clinical conditions, or participants potentially at risk of noncompliance to study procedures.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 8 Years to 34 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2028-03-06 (Estimated); Study Completion 2028-03-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Stage 3 Type 1 Diabetes based on American Diabetes Association criteria | From baseline up to Week 104
Change from baseline in area under the curve (AUC) of C-peptide | From baseline up to Week 104
Change from baseline in endogenous insulin | From baseline up to Week 104
Number of participants with TEAEs, SAEs, AEs leading to permanent study intervention- or study discontinuation; AEs of special interest; number of participants with clinically significant changes in vital signs, ECG, and/or safety laboratory test | Throughout the study, approximately 756 days
  TEAE: treatment-emerged adverse event; SAE: serious adverse event; AE: adverse event

SECONDARY OUTCOMES:
Change from baseline in fasting plasma glucose (FPG) from an oral glucose tolerance test | From baseline up to Week 104
Change from baseline in 2-hour plasma glucose from an oral glucose tolerance test | From baseline up to Week 104
Change from baseline of hemoglobin A1c (HbA1c) | From baseline up to Week 104
Serum concentration of teplizumab | From Day 1 to Day 28
CD3 receptor occupancy | From baseline to Day 28
Number of participants with anti-drug antibodies | From baseline up to Week 104
Number of participants with neutralizing antibodies | From baseline up to Week 104

CONTACTS AND LOCATIONS:
Locations (11):
- Japan (11):
  - Investigational Site Number : 3920015, Ichikawa, Chiba
  - Investigational Site Number : 3920006, Sapporo, Hokkaido
  - Investigational Site Number : 3920018, Kobe, Hyōgo
  - Investigational Site Number : 3920007, Yahaba, Iwate
  - Investigational Site Number : 3920019, Yokohama, Kanagawa
  - Investigational Site Number : 3920001, Iruma, Saitama
  - Investigational Site Number : 3920010, Chūō, Yamanashi
  - Investigational Site Number : 3920017, Fukuoka
  - Investigational Site Number : 3920016, Kyoto
  - Investigational Site Number : 3920004, Osaka
  - Investigational Site Number : 3920020, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: ACT18487 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=26396&tenant=MT_SNY_9011